CLINICAL TRIAL: NCT04646837
Title: Mechanism of Response to IMFINZI Neoadjuvant Therapy in Non-small Cell Lung Cancer Patients Based on Multiple-omics Models
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-IMFINZI-001
Record Dates: First submitted 2020-11-10; First posted 2020-11-30 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: neoadjuvant immunotherapy; IMFINZI; multiple-omics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Durvalumab 1000 mg IV Q3W + Paclitaxel 200mg/m2 + Carboplatin AUC 6 IV Q3W in resectable stage IB-IIIA NSCLC adult patients followed by adjuvant treatment for 1 year with Durvalumab 1000 mg IV Q3W for 4 months and Durvalumab 15000mg Q4W for 8 months
  Interventions: Drug: Durvalumab; Drug: Albumin Paclitaxel; Drug: Carboplatin/Cisplatin

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1000 mg IV Q3W for 2 cycle + Followed by adjuvant treatment for 1 year with Durvalumab 1000 mg IV Q3W for 4 months and Durvalumab 1500mg Q4W for 8 months
  Other Names: IMFINZI
Drug: Albumin Paclitaxel — Albumin Paclitaxel 200-260 mg, depending on the patient's physical condition, for 2 cycle
Drug: Carboplatin/Cisplatin — Carboplatin AUC 6 IV Q3W or Cisplatin 80mg/㎡ for 2 cycle

SUMMARY:
A single-center prospective exploratory single-arm neoadjuvant therapy study, based on a prospective cohort study, according to patients' blood and tumor samples before and after neoadjuvant treatment, WES, GEP gene expression profiling, TCR sequencing and ctDNA dynamic monitoring were used to explore the intratumoral immune consequences of PD-1 monoclonal antibody administration and identify potential Response biomarker.

DETAILED DESCRIPTION:
To explore the safety and immunobiological effects of 2 cycles of duvalumab combined with albumin paclitaxel + cisplatin/carboplatin for patients with stage IB-IIIA non-small cell lung cancer; use whole exome sequencing , GEP gene expression profile detection based on NanoString platform and other methods to predict the efficacy of IMFINZI neoadjuvant therapy, looking for potential biomarkers; study the impact of neoadjuvant therapy of I drug on the tumor microenvironment at multiple levels such as genome, transcriptome, PD-1/PD-L1 protein transcription and expression, T cell TCR immune groupthe library and T cell subsets, and provide comprehensive exploratory research evidence for finding the biomarker for the neoadjuvant anti-PD-L1 therapy of lung cancer .

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Male or female (no fertility requirement)
* Meet NCCN lung cancer diagnostic criteria
* No radical mastectomy, radiotherapy, chemotherapy, targeted therapy and immunotherapy
* Resectable stage Ib-IIIa non-small cell lung cancer (NSCLC) patients confirmed by imaging and biopsy; clear lung histopathological sample results have been obtained during screening, and all molecular biological tests can be completed.
* Patients without serious comorbidities, including but not limited to basic cardiovascular and cerebrovascular diseases, and patients whose clinical conditions allow to tolerate thoracic surgery
* Female and male subjects of childbearing age must use appropriate contraceptive measures during the study period and 6 months after the last study medication. Female subjects of childbearing age must have a negative pregnancy test
* Pathologically confirmed as lung adenocarcinoma or squamous cell carcinoma

Exclusion Criteria:

* Patients with unstable vital signs, need vasoactive drugs, or need intensive care unit (ICU) support
* Patients with active infections (including infections such as bacteria, fungi, viruses, tuberculosis, and various types of hepatitis) within 3 months before the first study medication
* Symptoms and signs of severe or uncontrolled liver, kidney, gastrointestinal, endocrine, lung, heart, neuropsychiatric, or brain disease
* Patients with a history of autoimmune diseases (inflammation or insufficiency of glands such as thyroid, pituitary, adrenal gland, etc., immunological diseases with positive autoantibodies)
* Is participating in other drug trials
* One month before the enrollment plan to receive immunotherapy, he had used any anti-systemic antibiotic therapy, hormone therapy, immunosuppressive therapy, etc.
* The pathology is small cell lung cancer or other neuroendocrine tumors or sarcomas, rare tumors or lung adenocarcinoma/squamous cell carcinoma containing the above components.
* The patient has a history of malignant tumors other than lung cancer
* Patients with sensitive gene mutations in EGFR (E19del/E21 L858R) and ALK (various types of fusion mutations)

Ages: 80 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
MPR | At the date of tumor assessment after surgery, estimated at approximately 24 weeks post-baseline
  Major pathologic response is defined as the presence of 10% or less of vital tumor cells in the sections of the primary lesion and/or mediastinal lymph nodes presenting focal microscopic disease after surgery

SECONDARY OUTCOMES:
Progression free survival | at 24 months from the first dose of neadjuvant treatment
  The progression free survival is the time until the patients disease progresses
Overall survival | at 3 years from the first dose of neoadjuvant treatment
  Time when the patient is still alive
Toxicity profile | from the first dose of neoadjuvant treatment until 90 days after the last dose of adjuvant treatment
  Toxicities caused by the drug during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No